CLINICAL TRIAL: NCT06336044
Title: "Clinical and Instrumental Evaluation of the Safety and Bio-revitalizing Effect on the Face of the Medical Device 'Volumizing Filler Based on Hyaluronic Acid and Recombinant Collagen'"
Brief Title: Pre-marketing Trial to Assess Safety and Efficacy of 'Volumizing Filler Based on Hyaluronic Acid and Recombinant Collagen'
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taumedika s.r.l. (Industry)
Collaborators: Nextrasearch S.r.l.s. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Taufiller/22
Record Dates: First submitted 2024-03-14; First posted 2024-03-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Wrinkle; Scar; Laxity; Skin
Keywords: hyaluronic acid; Collagen; Filler; Wrinkles
MeSH Terms: conditions — Cicatrix; Cutis Laxa

STUDY DESIGN:
Intervention Model Description: 20 patients for face and 20 for lips will undergo skin characterists measurments at time 0 at +4weeks and at +16 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face treatment (Experimental): Patients treated for face needs with Karisma micro injections
  Interventions: Device: Karisma
- Lips treatment (Experimental): Patients treated for face needs with Karisma microinjections
  Interventions: Device: Karisma

INTERVENTIONS:
Device: Karisma — Intradermal injection
  Other Names: Karisma filler

SUMMARY:
Study to validate the safety and efficacy of the Hyaluronic Acid +Collagen filler 40 patients will undergo through 3 visits one to asses the health and apply the filler one after 4 weeks to check the results one after 16 weeks for the final check and results validation Safety assessed with analysis of the Adverse Events

DETAILED DESCRIPTION:
The patients chosen with facial laxity characteristics, at the first visit will be assessed and will receive the treatment (microinjections) in the cheekbone area, over the lips and in the marionette lines. After 4 weeks the first visit will assess the change of the tissutal structure with non invasive measurements.

ELIGIBILITY:
Inclusion Criteria:

* all sexes
* caucasic
* 18 to 70 years
* non smoker

Exclusion Criteria:

* Pregnancy
* milking
* smoker
* alcohol or drugs abuse
* change of BMI during the study
* previous facial surgery, implants, permanent treatments
* sensitivity to the product
* dermatological difficult frame
* health weakness
* treated with anticoagulants, antihistaminics, corticosteroids, antidepressants and other drugs impacting on the results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety: no adverse events | 16 weeks
  test the safety of the device evaluating any potential adverse event
Efficacy: change of wrinkles and scars | 16 weeks
  test the efficacy of the device measuring the skin surface using GAIS (Global Aesthetic Improvement Scale) scale
Efficacy: change of wrinkles and scars | 16 weeks
  test the efficacy of the device measuring the skin surface using Facial Volume Loss Scale (FVLS)
Efficacy: change of wrinkles and scars | 16 weeks
  test the efficacy of the device measuring the skin surface evaluating the face volume
Efficacy: change of wrinkles and scars | 16 weeks
  test the efficacy of the device measuring the skin surface with skin hydratation measurement

SECONDARY OUTCOMES:
Duration of the efficacy | 16 weeks
  measure the duration of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Gasparetto, MD, Study Director — Nextrasearch S.r.l.s.
Locations (1):
- Ospedale Tor Vergata, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
Not foreseen